CLINICAL TRIAL: NCT04568174
Title: First in Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of PPSGG (PN-1007) in Anti-MAG Neuropathy Patients
Brief Title: First in Human Study to Test the Safety and Preliminary Efficacy of PPSGG in Patients With Anti-MAG Neuropathy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Data don't support further development
Sponsor: Polyneuron Pharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PN-1007-001
Record Dates: First submitted 2020-09-08; First posted 2020-09-29 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Anti-MAG Neuropathy
Keywords: peripheral neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Single Group in SAD and parallel in MAD
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The SAD phase is open label and MAD is randomized, dose escalation, double blind (patient and investigator blinded), placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPSGG (Active Comparator): sterile liquid, one 1-hour infusion in SAD and multiple infusions in MAD. In SAD multiple cohorts being tested. Dosage and regime in MAD to be defined based on SAD outcome.
  Interventions: Drug: PPSGG
- Placebo (Placebo Comparator): standard PBS solution, pH 7.4, composed of disodium hydrogen phosphate dodecahydrate, potassium dihydrogen phosphate, sodium chloride, and water for injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PPSGG — an antibody scavenger of pathogenic anti-MAG immunoglobulin M (IgM) autoantibodies
  Other Names: PN-1007
  Arms: PPSGG
Drug: Placebo — A standard PBS solution, pH 7.4, composed of disodium hydrogen phosphate dodecahydrate, potassium dihydrogen phosphate, sodium chloride, and water for injection
  Arms: Placebo

SUMMARY:
In this study, the new drug called PPSGG (PN-1007) will be tested. Preliminary studies conducted in animals suggest PPSGG (PN-1007) might be a good treatment for reducing levels of anti-MAG antibodies in patients with anti-MAG neuropathy.

This is the first research of PPSGG (PN-1007) in people and its main purpose is to test its safety and acceptability in patients. In this study it will be examined how the drug is changed by and removed from the body and checked for signs that the drug may be truly effective against anti-MAG neuropathy. PPSGG (PN-1007) will be tested at several different doses.

DETAILED DESCRIPTION:
PPSGG (PN-1007) is intended to bind anti-MAG IgM autoantibodies, the underlying cause of anti-MAG neuropathy, in a highly selective manner, resulting in their neutralization and removal from the circulation. This allows specific targeting of anti-MAG IgM in the circulation and circumvents unspecific immunosuppression associated with current treatment strategies.

This is a Phase I/IIa, First in Human (FiH), multicenter, single and multiple ascending dose escalation trial of PPSGG (PN-1007), an antibody scavenger of pathogenic anti-MAG immunoglobulin M (IgM) autoantibodies for treatment of anti-MAG neuropathy. The aim of the study is to assess the safety and tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of PPSGG (PN-1007) in a SAD and a MAD phase in an adaptive trial in anti-MAG neuropathy patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of monoclonal IgM associated with MGUS with anti-MAG activity (titer of > 10'000 BTU) and demyelinating neuropathy defined by electrophysiological criteria according to EFNS/PNS PDN guideline, 2010.
* Clear clinical signs of disability
* Adequate hepatic and renal function

Exclusion Criteria:

* Patients with total serum IgM levels >30 g.
* Hematological malignancy, prior malignancy of any organ system (except BCC)
* Prior immunosuppression: No IVIG in previous 3 months, no previous cyclophosphamide or biologicals in prior 6 months.
* Other neurological, neuromuscular, rheumatologic or orthopedic condition with significant impact on the capabilities of walk preventing evaluation of neurological scores

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) | 1 month
  All AEs will be recorded, whether considered minor or serious, drug-related or not
anti-drug-antibodies ADA | 1 month in SAD
  Potential ADAs (immunogenicity) resulting from exposure of patients to PPSGG (PN-1007) will be measured by ELISA

SECONDARY OUTCOMES:
Tmax | Day 1 to Day 42
  Time of peak concentration of PPSGG (PN-1007)
Cmax | Day 1 to Day 42
  Maximum Plasma Concentration of PPSGG (PN-1007)
AUCinf | Day 1 to Day 42
  Area under the plasma concentration versus time curve from zero to infinity of PPSGG (PN-1007)
t1/2 | Day 1 to Day 42
  Terminal half life of PPSGG (PN-1007)
Pharmacodynamic | up to Day 28
  Change in anti-MAG Buhlmann titer from baseline measured by ELISA
Change From Baseline in ONLS | up to Day 150 in MAD
  Overall Neuropathy Limitations Scale measures limitations in the everyday activities of the upper and lower limbs

CONTACTS AND LOCATIONS:
Overall Officials: Hedvika Lazar, Study Chair — Polyneuron Pharmaceuticals AG
Locations (7):
- France (3):
  - Service de Neurologie Centre de Référence Neuropathies Périphériques Rares, CHU Limoges, Limoges
  - Referral centre for neuromuscular diseases and ALS, hôpital La Timone, Marseille
  - Département de Neurologie Pôle Neurosciences Centre de Référence des Neuropathies Amyloïdes Familiales et autres Neuropathies Périphériques Rares Centre Hospitalier Universitaire de Bicêtre, Paris
- UMC Utrecht Cancer Center, Utrecht, Netherlands
- Barcelona, Barcelona, Spain
- Lausanne, Lausanne, Switzerland
- National hospital for neurology and neurosurgery, Queen London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No